CLINICAL TRIAL: NCT03510000
Title: Alleviating Carbohydrate-Counting Burden in Type 1 Diabetes Using Artificial Pancreas and Sodium Glucose-Linked Transporter 2 Inhibition: A Randomized Open-Label Crossover Trial.
Brief Title: Alleviating Carbohydrate-Counting Burden in T1DM Using Artificial Pancreas and Empagliflozin
Acronym: CLASS15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: Canadian Diabetes Association (Other); Institut de Recherches Cliniques de Montreal (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLASS15
Record Dates: First submitted 2018-01-24; First posted 2018-04-27 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Type1diabetes
Keywords: T1DM; artificial pancreas; insulin pump; empagliflozin; SGLT2 inhibitor; carbohydrate counting
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main arm (Experimental): Single arm open-label cross-over study with random order of SGLT-2 inhibitor intervention (Empagliflozin 25mg po qd), in which each cross-over phase includes different meal strategies (carbohydrate counting, meal announcement, no meal announcement) on separate days in the setting of single hormone artificial pancreas
  Interventions: Drug: Empagliflozin 25mg; Device: Single hormone artificial pancreas; Behavioral: Meal strategies

INTERVENTIONS:
Drug: Empagliflozin 25mg — Individuals will test insulin dosing during different meal strategies (carbohydrate counting, plain meal announcement, no meal announcement) in a setting of the single hormone artificial pancreas with or without SGLT2 inhibitor (empagliflozin) addition. After starting the empagliflozin therapy, there will be 1-2 weeks long therapy optimization period and afterwards meal strategies will be administered. Randomization will be used to determine whether participant will start meal strategies on empagliflozin or without empagliflozin, cross-over design enables all participants to undergo all combination of approaches.
Device: Single hormone artificial pancreas — Single hormone artificial pancreas will be used as a baseline background intervention standardizing the delivery and dosing of insulin. Artificial pancreas (insulin pump, continuous glucose monitoring device and dosing-suggestion algorithm) will be used by all participants on days when meal strategy intervention will be performed.
Behavioral: Meal strategies — Participants will use different approaches (strategies) to insulin dose estimation for ingested carbohydrates on study days. Goal of these various strategies is to recognize magnitude of empagliflozin effect in situations when artificial pancreas algorithm is working with information of different accuracy. Individual meal approach strategies include carbohydrate counting, meal size announcement and no meal announcement. The exception will be combination of no empagliflozin and no meal announcement, which didn't result in sufficient glucose control in previous trials therefore will not be repeated in a current trial. Meal approach strategies will occur on separate days- 5 days in total each day using one meal strategy for all meals during the day.

SUMMARY:
One of the challenges in the design of the artificial pancreas (AP) is preventing postprandial hyperglycemia. Beyond algorithmic solutions, one countermeasure to postprandial hyperglycemia that may enhance performance of the AP is the use of adjunctive-to-insulin medications such as those in the Sodium Glucose-Linked Transporter 2 inhibitor class. This study evaluates whether use of oral empagliflozin on the background of single-hormone AP can improve postprandial blood glucose control. The investigators will test this hypothesis in a cross-over trial design by comparing open-label empagliflozin versus placebo in the setting of AP on separate study days that involve carbohydrate counting, simple meal announcement and no meal announcement strategies.

DETAILED DESCRIPTION:
Empagliflozin is a novel anti-diabetic medication and has been approved in Canada. The labelled indication for use of empagliflozin in clinical practice is as an adjunct therapy to diet and exercise to improve glycemic control in adult patients with type 2 diabetes. The investigators are proposing to use the medication as an adjunct anti-diabetic therapy in individuals with type 1 diabetes and would like to examine whether empagliflozin can alleviate need for carb-counting by eliminating post-prandial hyperglycemia in a setting of an artificial pancreas (AP).

The study is designed as a randomized open-label, crossover non-inferiority trial comparing empagliflozin 25 mg oral daily in the setting of the single-hormone AP to single-hormone AP without empagliflozin in adults with type 1 diabetes. The duration of the study for each of the participants is about 3-9 weeks and during this time three different meal announcement strategies for AP will be used, on and off empagliflozin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year.
2. Use of insulin pump therapy for at least 3 months.
3. HbA1c ≤ 10%.
4. Women of childbearing potential must agree to use adequate birth control during participation in the study

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy.
2. Recent acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. History of pheochromocytoma or insulinoma
4. Use of loop diuretics, anticholinergic drugs, beta-blockers at high dose, glucocorticoids (except low stable dose and inhaled steroids), chronic acetaminophen treatment, chronic warfarin treatment
5. Use of non-insulin adjunct anti-hyperglycaemic drug (e.g. metformin, glucagon-like peptide analogues, etc.).
6. Ongoing or planned pregnancy or breastfeeding.
7. Recent severe hypoglycemic episode prior to enrollment
8. Recent diabetic ketoacidosis prior to enrollment
9. Recent history of genital or urinary infection prior to enrollment
10. History of lower limb amputation and recent history of leg or foot infection or wound
11. Anticipating a significant change in exercise regimen between initiations of two intervention blocks (i.e. starting or stopping an organized sport).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Comparison of mean glucose levels between artificial pancreas (AP) with empagliflozin with no-meal announcement meal approach strategy and AP without empagliflozin with carb-counting meal approach strategy. | After completing 5 meal interventions (3-9 weeks)
  Non-inferiority comparison of mean 14-hour glucose level obtained by continuous glucose monitoring between i) the AP with empagliflozin with no meal-announcement and ii) the AP with quantitative carbohydrate-counting without empagliflozin.
Comparison of mean glucose levels between AP with empagliflozin with simple meal announcement strategy and AP without empagliflozin with carb-counting. | After completing 5 meal interventions (3-9 weeks)
  If there is a significant difference in the previous non-inferiority comparison, the following conditional primary comparison will be conducted:
  Non-inferiority comparison of mean 14-hour sensor glucose level obtained by continuous glucose monitoring between i) the AP with empagliflozin with simple meal-announcement and ii) the AP with quantitative carbohydrate-counting without empagliflozin.

SECONDARY OUTCOMES:
Time spent in hypoglycemia | After completing 5 meal interventions (3-9 weeks)
  Percentage of time spent in the following glucose sensor levels:
  1. Between 3.9 and 10.0 mmol/l
  2. Between 3.9 and 7.8 mmol/l
  3. Above 7.8 mmol/l
  4. Above 10.0 mmol/l
  5. Above 13.9 mmol/l
  6. Below 3.9 mmol/l
  7. Below 3.3 mmol/l
  8. Below 2.8 mmol/l.
Number of hypoglycemic events below 3.3 mmol/L | After completing 5 meal interventions (3-9 weeks)
  Number of hypoglycemic events (> 20 minutes) below 3.3 mmol/L based on continuous glucose monitoring sensor glucose level values.
Number of clinically remarkable hypoglycemic events | After completing 5 meal interventions (3-9 weeks)
  Number of symptomatic hypoglycemic events below 4.0 mmol/l or below 3.5 mmol/l without symptoms.
Number of treated hypoglycemic events | After completing 5 meal interventions (3-9 weeks)
  Number of hypoglycemic events or events perceived as hypoglycemia which prompt treatment by glucose or glucagon or overriding AP insulin dosing algorithm suggestion or by administering the regular meal earlier than planned.
Mean continuous glucose monitoring (CGM) glucose level | After completing 5 meal interventions (3-9 weeks)
  Comparison of mean CGM glucose levels between different meal interventions on and off empagliflozin.
Standard deviation of glucose levels | After completing 5 meal interventions (3-9 weeks)
  Comparison of values obtained from CGM on different meal intervention days.
Coefficient of variation of glucose levels | After completing 5 meal interventions (3-9 weeks)
  Comparison of values obtained from CGM on different meal intervention days.
Total insulin delivery | After completing 5 meal interventions (3-9 weeks)
  Comparison of total insulin delivered by AP on different meal intervention days.
Morning capillary ketone concentration | After completing 5 meal interventions (3-9 weeks)
  Safety outcome to assess risk of Empagliflozin related most serious side effect-diabetic ketoacidosis. Evaluated will be all days of study participation (i.e.not only meal intervention days)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Perkins, MD, Principal Investigator — Samuel Lunenfeld Research Institute, TGRI
Locations (3):
- Canada (3):
  - Sinai Health System, Toronto, Ontario
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No